CLINICAL TRIAL: NCT04162288
Title: RCT Protocol for Evaluating an Online Training Program on Shared Decision-making About Screening for Down Syndrome
Brief Title: Evaluating an Online Training Program on Shared Decision-making in Prenatal Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Genome Quebec (Other); Genome Canada (Other); CERSSPL (Unknown)
Responsible Party: Principal Investigator, France Legare, Principal investigator, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MP-20-2019-4571
Record Dates: First submitted 2019-08-22; First posted 2019-11-14 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Shared Decision Making
Keywords: Shared Decision Making; Decision aid; Nurse; Online Training

STUDY DESIGN:
Intervention Model Description: This is a multi-center, two-arm, controlled trial (RCT). Thirty-six participants will be randomly allocated to either 1) an experimental group that is exposed to our complete 3 hours online training program intervention (n = 18) or 2) a control group that is exposed to an intervention which will be a 3 hours online training program focused on prenatal screening.
Who Masked: Participant, Care Provider, Investigator
Masking Description: When a participant is randomised to the trial, the private firm will assign a trial group following a pre-selected list of randomisation (given by the private firm). The employee of the private firm will be the one non-blinded in our study, by giving participant access to one of the formation. The ''Care Provider'' is not present in this study; in fact, all interactions are via the private firm and is directed towards an online-intervention. A randomisation list will be kept by the private firm and send to the research team after the data analysis. The Investigator are blinded also by the randomisation process. There is no officially Outcomes Assessor, because the outcomes of interest are self-reported (intention of using a DA) or pre-measured (for example; with the knowledge test, rightful answer are already known).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online training on SDM in prenatal screening (Experimental)
  Interventions: Other: Online Training - Shared Decision Making in Prenatal Screening
- Online training on prenatal screening (Placebo Comparator)
  Interventions: Other: Online Training - Online Training on Prenatal Screening

INTERVENTIONS:
Other: Online Training - Shared Decision Making in Prenatal Screening — TThe intervention consisted of an online self-study training program lasting 3 hours which aims to engage SDM in a prenatal screening context. The training was divided into four main modules: 1)SDM, 2)DS prenatal screening, 3)Decision aid and 4)Communication between healthcare professionals and patients. In each module, the targeted learning objectives and the work to be carried out (e.g. readings to be made, video to be viewed, evaluation to be carried out, etc.) are presented. Various teaching methods and medias are used during this training: videos, interviews, narrated capsule, readings, links to scientific articles and complementary websites. Videos are done with experts on SDM, ethics of prenatal testing. A simulation in the end is done to put participants in context of an actual consultation with a pregnant woman and her partner. This training was designed to adapt to the learning pace of the user, is hosted on University Laval platform and needs an identification code to enter.
  Arms: Online training on SDM in prenatal screening
Other: Online Training - Online Training on Prenatal Screening — The control intervention consisted of an online self-study training program lasting 3 hours which aims to provides knowledge for prenatal screening. The training has four main modules: 1)Context and history of prenatal screening(new), 2)DS prenatal screening(existing), 3)Consent in prenatal screening(new) and 4)Communication between healthcare professionals and patients(existing). In each module, the targeted learning objectives and the work to be carried out are presented. Various teaching methods and medias are used during this training: videos, interviews, narrated capsule, readings, links to scientific articles and complementary websites. Videos are done with experts on SDM, ethics of prenatal testing. For the 2 new modules, narrated capsules and reports have replaced videos of experts. There is no simulation at the end. This training was designed to adapt to the learning pace of the user, is hosted on University Laval platform and needs an identification code to enter.
  Arms: Online training on prenatal screening

SUMMARY:
The investigators aim to evaluate an online training program on shared decision making within the prenatal context. The main outcome is intention on using a decision aid in prenatal screening consultation and study population is nurses. Secondary outcomes are; knowledge acquisition, acceptability of the formation and perceived usefulness. The investigators hypothesise that this web-based SDM training program developed for the prenatal screening of Down Syndrome will significantly increase nurses' intentions to use the decision aid in their clinical practice with pregnant women and their partner.

DETAILED DESCRIPTION:
Pregnant women have difficulty choosing among the wide variety of prenatal screening options available. To help pregnant women and their partners make informed decisions based on their values, needs and preferences, a decision aid (DA) has been developped and online shared decision-making (SDM) training program for health professionals has been created to support the use of this DA and give health care professionals key elements on SDM. The decision aid was found relevant and acceptable to pregnant women and their partners; the relevance and acceptability of the online SDM training program aren't evaluated yet. This study aim to assess the intention on using a DA after taking the online training program, to evaluate knowledge acquisition and to assess the program's acceptability and perceived usefulness. This is a multi-center, two-arm, controlled trial (RCT). Thirty-six participants will be randomly allocated to either 1) an experimental group that is exposed to the investigator's complete 3 hours online training program intervention (n = 18) or 2) a control group that is exposed to an intervention which will be a 3 hours online training program focused on prenatal screening alone.

ELIGIBILITY:
Inclusion Criteria:

* Be a certified nurse
* Be involved in supporting prenatal screening decision-making or involved in prenatal screening processes in the province of Quebec;
* Speak and write in French
* Being in active practice within the last year.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change of intention to use a decision aid after completing the online training program on SDM in prenatal screening | The intention will be measured initially before accessing the formation. After the formation completed (duration is variable), the participant will have access to the questionnaire once again in a delay of 24-72 hours.
  Nurses intention of using a decision aid for prenatal screening in clinical practice is the primary outcome. To be measured, the CPD (Continuing professional development) reaction questionnaire will be used. This questionaire scores on 5 constructs; intention, social influence, beliefs about capabilities, moral norm and beliefs about consequences and has 12 questions. The constructs intention will be targeted, however the others constructs will be also evaluated for their potential on predicting behavior of health professionals. It is a self-reported questionnaire. The use of decision aid has been chosen as an outcome become it is a main component of SDM itself and of the training. The score is on a scale from 1 to 7 (Likert type), which 1 is the minimum and 7 the maximum value (except one question that has a 5 intervals of pourcentage, that will be adjusted on 7 items scale in the analysis). The higher score means better outcome.

SECONDARY OUTCOMES:
Knowledge on aspects surrounding prenatal screening and SDM | After the formation completed (duration is variable), the participant will have access to the questionnaire in a delay of 24-72 hours.
  A newly designed and self-reported questionnaire consisting of 20 questions, reviewed by an SDM expert and a pedagogical advisor, explore knowledge on; Down Syndrome (2 questions), prenatal screening (7 questions), SDM (7 questions) and ethic (4 questions). There is 2 true-false questions and the other ones are multiple choices questions. Each question has the same ponderation, which is 5% on a total score of 100%. There is only one right answer to each question. There is no negative correction. The higher score means better outcome (acquisition of knowledge). The title of this questionnaire is: "Knowledge".
Satisfaction with training: self-reported questionnaire | After the formation completed (duration is variable), the participant will have access to the questionnaire in a delay of 24-72 hours.
  Satisfaction will be addressed on the content, trainers and overall satisfaction. For evaluating these kinds of satisfaction, a pre-existing self-reported questionnaire created by Schmidt (2007) will be used. The score is on a scale from 1 to 5 (Likert type), which 1 is the minimum and 5 the maximum value. The higher score means better outcome. The title of this section is :"Satisfaction" and it has two sections; "Satisfaction within the training content" and "Satisfaction with the training contributors".
Acceptability of the training: self-reported questionnaire | After the formation completed (duration is variable), the participant will have access to the questionnaire in a delay of 24-72 hours.
  Acceptability is evaluated by looking at the comprehensibility, the amount of information , the quality of information, the format chosen of the training and it is based on a pre-existing self-reported questionnaire done by Kasper and al. (2017). The score is on a scale from 1 to 5 (Likert type), which 1 is the minimum and 5 the maximum value. The higher score means better outcome. The title of this questionnaire is "Training acceptability".
Perceived usefulness | After the formation completed (duration is variable), the participant will have access to the questionnaire in a delay of 24-72 hours.
  Usefulness is declined in terms of work responsibilities, relevance of topics to career development, relevance of topics in relation to individual learning needs, consistency with declared objectives, balance between theory and practice and it is based on a self-reported questionnaire by Giangreco, Sebastiano and Peccei (2009). The score is on a scale from 1 to 5 (Likert type), which 1 is the minimum and 5 the maximum value. The higher score means better outcome. The title of this questionnaire is "Perceived usefulness of the formation".

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, PhD, Principal Investigator — VITAM - Centre de recherche en santé durable
Locations (1):
- Leger, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legare F, Witteman HO. Shared decision making: examining key elements and barriers to adoption into routine clinical practice. Health Aff (Millwood). 2013 Feb;32(2):276-84. doi: 10.1377/hlthaff.2012.1078. PMID 23381520
- [Background] Moulton B, Collins PA, Burns-Cox N, Coulter A. From informed consent to informed request: do we need a new gold standard? J R Soc Med. 2013 Oct;106(10):391-4. doi: 10.1177/0141076813490686. Epub 2013 Jun 6. No abstract available. PMID 23759895
- [Background] Gray M, Jani A. Promoting Triple Value Healthcare in Countries with Universal Healthcare. Healthc Pap. 2016;15(3):42-8. PMID 27009586
- [Background] Shay LA, Lafata JE. Where is the evidence? A systematic review of shared decision making and patient outcomes. Med Decis Making. 2015 Jan;35(1):114-31. doi: 10.1177/0272989X14551638. Epub 2014 Oct 28. PMID 25351843
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Legare F, Stacey D, Turcotte S, Cossi MJ, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2014 Sep 15;(9):CD006732. doi: 10.1002/14651858.CD006732.pub3. PMID 25222632
- [Background] Legare F, Adekpedjou R, Stacey D, Turcotte S, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for increasing the use of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2018 Jul 19;7(7):CD006732. doi: 10.1002/14651858.CD006732.pub4. PMID 30025154
- [Background] Legare F, St-Jacques S, Gagnon S, Njoya M, Brisson M, Fremont P, Rousseau F. Prenatal screening for Down syndrome: a survey of willingness in women and family physicians to engage in shared decision-making. Prenat Diagn. 2011 Apr;31(4):319-26. doi: 10.1002/pd.2624. Epub 2011 Jan 26. PMID 21268046
- [Background] St-Jacques S, Grenier S, Charland M, Forest JC, Rousseau F, Legare F. Decisional needs assessment regarding Down syndrome prenatal testing: a systematic review of the perceptions of women, their partners and health professionals. Prenat Diagn. 2008 Dec;28(13):1183-203. doi: 10.1002/pd.2059. PMID 19097031
- [Background] Couet N, Desroches S, Robitaille H, Vaillancourt H, Leblanc A, Turcotte S, Elwyn G, Legare F. Assessments of the extent to which health-care providers involve patients in decision making: a systematic review of studies using the OPTION instrument. Health Expect. 2015 Aug;18(4):542-61. doi: 10.1111/hex.12054. Epub 2013 Mar 4. PMID 23451939
- [Background] Legare F, O'Connor AC, Graham I, Saucier D, Cote L, Cauchon M, Pare L. Supporting patients facing difficult health care decisions: use of the Ottawa Decision Support Framework. Can Fam Physician. 2006 Apr;52(4):476-7. PMID 17327891
- [Background] Legare F, Ratte S, Gravel K, Graham ID. Barriers and facilitators to implementing shared decision-making in clinical practice: update of a systematic review of health professionals' perceptions. Patient Educ Couns. 2008 Dec;73(3):526-35. doi: 10.1016/j.pec.2008.07.018. Epub 2008 Aug 26. PMID 18752915
- [Background] Stacey D, Hill S, McCaffery K, Boland L, Lewis KB, Horvat L. Shared Decision Making Interventions: Theoretical and Empirical Evidence with Implications for Health Literacy. Stud Health Technol Inform. 2017;240:263-283. PMID 28972523
- [Background] Legare F, Stacey D, Briere N, Fraser K, Desroches S, Dumont S, Sales A, Puma C, Aube D. Healthcare providers' intentions to engage in an interprofessional approach to shared decision-making in home care programs: a mixed methods study. J Interprof Care. 2013 May;27(3):214-22. doi: 10.3109/13561820.2013.763777. Epub 2013 Feb 8. PMID 23394265
- [Background] Leiva Portocarrero ME, Garvelink MM, Becerra Perez MM, Giguere A, Robitaille H, Wilson BJ, Rousseau F, Legare F. Decision aids that support decisions about prenatal testing for Down syndrome: an environmental scan. BMC Med Inform Decis Mak. 2015 Sep 24;15:76. doi: 10.1186/s12911-015-0199-6. PMID 26404088
- [Background] Delanoe A, Lepine J, Turcotte S, Leiva Portocarrero ME, Robitaille H, Giguere AM, Wilson BJ, Witteman HO, Levesque I, Guillaumie L, Legare F. Role of Psychosocial Factors and Health Literacy in Pregnant Women's Intention to Use a Decision Aid for Down Syndrome Screening: A Theory-Based Web Survey. J Med Internet Res. 2016 Oct 28;18(10):e283. doi: 10.2196/jmir.6362. PMID 27793792
- [Background] Delanoe A, Lepine J, Leiva Portocarrero ME, Robitaille H, Turcotte S, Levesque I, Wilson BJ, Giguere AM, Legare F. Health literacy in pregnant women facing prenatal screening may explain their intention to use a patient decision aid: a short report. BMC Res Notes. 2016 Jul 11;9:339. doi: 10.1186/s13104-016-2141-0. PMID 27401163
- [Background] Portocarrero ME, Giguere AM, Lepine J, Garvelink MM, Robitaille H, Delanoe A, Levesque I, Wilson BJ, Rousseau F, Legare F. Use of a patient decision aid for prenatal screening for Down syndrome: what do pregnant women say? BMC Pregnancy Childbirth. 2017 Mar 20;17(1):90. doi: 10.1186/s12884-017-1273-0. PMID 28320334
- [Background] WHO. Nine steps for developing a scaling-up strategy Geneva: World Health Organization; 2010. Available from: http://www.who.int/iris/handle/10665/44432.
- [Background] Legare F, Borduas F, Freitas A, Jacques A, Godin G, Luconi F, Grimshaw J; CPD-KT team. Development of a simple 12-item theory-based instrument to assess the impact of continuing professional development on clinical behavioral intentions. PLoS One. 2014 Mar 18;9(3):e91013. doi: 10.1371/journal.pone.0091013. eCollection 2014. PMID 24643173
- [Background] Schmidt SW. The relationship between satisfaction with workplace training and overall job satisfaction. Human Resource Development Quarterly. 2007;18(4):481-98.
- [Background] Kasper J, Liethmann K, Heesen C, Reissmann DR, Geiger F. Training doctors briefly and in situ to involve their patients in making medical decisions-Preliminary testing of a newly developed module. Health Expect. 2017 Dec;20(6):1254-1263. doi: 10.1111/hex.12565. Epub 2017 May 18. PMID 28521082
- [Background] Giangreco A, Sebastiano A, Peccei R. Trainees' reactions to training: an analysis of the factors affecting overall satisfaction with training. The international journal of human resource management. 2009;20(1):96-111.
- [Background] Kirkpatrick D, Kirkpatrick J. Evaluating Training Programs: The four levels. San Francisco, CA, USA: Berret-Koehler Publishers, Inc.; 2009
- [Background] Abbasgholizadeh Rahimi S, Lepine J, Croteau J, Robitaille H, Giguere AM, Wilson BJ, Rousseau F, Levesque I, Legare F. Psychosocial Factors of Health Professionals' Intention to Use a Decision Aid for Down Syndrome Screening: Cross-Sectional Quantitative Study. J Med Internet Res. 2018 Apr 25;20(4):e114. doi: 10.2196/jmir.9036. PMID 29695369
- [Derived] Poulin Herron A, Agbadje TT, Cote M, Djade CD, Roch G, Rousseau F, Legare F. Web-Based Training for Nurses on Shared Decision Making and Prenatal Screening for Down Syndrome: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Oct 29;9(10):e17878. doi: 10.2196/17878. PMID 33118955